CLINICAL TRIAL: NCT05028855
Title: Cerebral Autoregulation in Patients With Symptomatic Cerebral Atherosclerotic Stenosis
Acronym: CASCAS
Status: Recruiting | Type: Observational
Sponsor: Yi Yang (Other)
Collaborators: Shenzhen Second People's Hospital (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The First Affiliated Hospital of University of South China (Other); Eighth Affiliated Hospital, Sun Yat-sen University (Other); The First Affiliated Hospital of Hebei North University (Other); Qilu Hospital of Shandong University (Other); The Affiliated Hospital of Qingdao University (Other); The Affiliated Hospital of Yanbian University (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: CASCAS
Record Dates: First submitted 2017-07-19; First posted 2021-08-31 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Cerebrovascular Stroke; Cerebral Artery Stenosis
Keywords: cerebral atherosclerotic stenosis; ischemic stroke; transient ischemic attack; cerebral autoregulation
MeSH Terms: conditions — Stroke; Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sCAS patients: Investigators plan to enroll 850 patients of symptomatic cerebral atherosclerotic stenosis (sCAS) for cerebral autoregulation assessment to explore the relationship between cerebral autoregulation (CA) and stroke recurrence, determine the threshold values of CA parameter for predicting stroke recurrence associated with particular stenosis.
  Interventions: Diagnostic Test: Cerebral autoregulation assessment

INTERVENTIONS:
Diagnostic Test: Cerebral autoregulation assessment — Cerebral autoregulation assessment will be conducted by specialized neurovascular ultrasound doctors during 0-3 and 10-30 days after stroke onset.The recorded data will be stored for further cerebral autoregulation analysis.

SUMMARY:
In this multi-center prospective observational study within a cohort of symptomatic cerebral atherosclerotic stenosis (sCAS) patients, 850 subjects were planed to be enrolled to explore the relationship between cerebral autoregulation (CA) and stroke recurrence, determine the threshold values of CA parameter for predicting stroke recurrence associated with particular stenosis.

DETAILED DESCRIPTION:
Ischemic stroke is a tremendous public health burden that seriously endangers the health of Chinese population symptomatic cerebral atherosclerotic stenosis (sCAS) is responsible for about 33-50% of ischemic stroke in China and highly associated with the risk of stroke recurrence.

Cerebral autoregulation (CA) is the main protective mechanism that modulates cerebral blood flow to satisfy regional cerebral perfusion demands despite of variations in arterial blood pressure (ABP). Thus, CA supposed to be particularly considered when choosing individual therapeutic strategy in sCAS patients. In clinical practice, applying transcranial Doppler combined with servo-controlled plethysmograph assessing CA has been proved a feasible method in cerebral atherosclerotic stenosis patients. Especially in those severe stenosis patients, CA is probably compromised in varying degrees, whereas whether and to what extent CA parameters have the capability to predict stroke recurrence has not been illustrated.

Thus, the aim of the study was to assess CA after acute ischemic stroke or transient ischemic attack within 2 years follow-up to explore the relationship between CA and stroke recurrence and determine the threshold values of CA parameter to predict stroke recurrence. CA measurement will be performed at 0-3 and 10-30 days after ischemic cerebrovascular events. Clinical information, neuroimaging data, biochemical examinations and follow-up information will be collected and recorded in case report form (CRF) once signing of informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 18 to 80, both genders
* Unilateral internal carotid artery (ICA) or M1 segment of middle cerebral artery (MCA) stenosis (rate of stenosis ranging from 50-99%)
* Acute ischemic cerebrovascular events (TIA or ischemic stroke) within cerebral stenotic artery supplying area
* Onset of disease <30 d before enrollment
* Modified Ranking Scale (mRS) ≤1 before stroke onset
* National Institutes of Health Stroke Scale (NIHSS) ≤20
* Sufficient bilateral temporal bone windows for insonation of the middle cerebral artery
* Be conscious, and able to cooperate with CA assessment
* Willing to participate and sign the informed consent

Exclusion Criteria:

* Vertebral artery (VA), basilar artery (BA), anterior cerebral artery (ACA), or posterior cerebral artery (PCA) stenosis; Bilateral internal carotid artery (ICA) or M1 segment of middle cerebral artery (MCA) stenosis(rate of stenosis ranging from 50-99%)
* Patients who have received or plan to undergo intravascular interventional treatment/endarterectomy
* Other intracranial diseases, including cerebral hemorrhage (primary or secondary), intracranial neoplasm, aneurysm, arteriovenous malformation, etc.
* Evidence for embolic stroke, such as atrial fibrillation, prosthetic valve surgery, and suspected endocarditis, etc.
* Arrhythmia, anemia and hyperthyroidism which may influence the stability of cerebral blood flow diagnosed by two physicians by electrocardiogram and laboratory tests.
* Dementia, severe anxiety, depression, and other mental diseases
* Malignant neoplasm and expected lifetime <2 years
* Enrolled in other clinical trails within 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of symptomatic cerebral atherosclerotic stenosis, were recruited according to Inclusion Criteria, mostly from the First Hospital of Jilin University, and partly from other hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2017-01-14 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Stroke recurrence rate | two years
  Ischemic cerebrovascular recurrence (TIA or ischemic stroke) within cerebral stenotic artery supplying area diagnosed by symptoms and imaging examinations.

SECONDARY OUTCOMES:
The index of cerebral autoregulation | within 30 days ischemic cerebrovascular events onset
  Phase difference, gain and coherence of symptomatic cerebral atherosclerotic stenosis patients within 30 days ischemic cerebrovascular events onset.
ischemic cerebrovascular recurrence rate | two years
  All ischemic cerebrovascular recurrence (TIA or ischemic stroke) within two years follow-up diagnosed by symptoms and imaging examinations.
The first onset time of composite endpoint events within 2 years | two years follow-up
  The composite endpoint events include fatal and nonfatal stroke (ischemic or hemorrhagic stroke), fatal and nonfatal myocardial infarction, transient ischemic attack (TIA) diagnosed by symptoms and imaging examinations.
mRS and Barthel score | two years
  The changes of mRS and Barthel score within 2 years
The first onset time of each individual part of composite endpoint events within 2 years | two years follow-up
  The first onset time of each individual part of composite endpoint events within 2 years
the NIHSS score | within 1 month
  The changes of NIHSS score from admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, MD, PhD, Study Chair — Neuroscience Center, Department of Neurology, The First Hospital of Jilin University
Locations (1):
- the First Hospital of Jilin University, Changchun, Jilin, China